CLINICAL TRIAL: NCT06620302
Title: DT2216 in Combination With Irinotecan for Children, Adolescents and Young Adults With Relapsed or Refractory Solid Tumors: A Phase I Study With Phase II Feasibility Cohort for Fibrolamellar Carcinoma
Brief Title: Testing the Addition of an Anti-cancer Drug, DT2216, to the Usual Chemotherapy Treatment for Relapsed or Refractory Solid Tumors and Fibrolamellar Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEPN2411; NCI-2024-06357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN2411 (Other: Pediatric Early Phase Clinical Trial Network); PEPN2411 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-07

CONDITIONS: Childhood Fibrolamellar Carcinoma; Recurrent Childhood Fibrolamellar Carcinoma; Recurrent Childhood Malignant Solid Neoplasm; Recurrent Fibrolamellar Carcinoma; Recurrent Malignant Solid Neoplasm; Refractory Childhood Fibrolamellar Carcinoma; Refractory Childhood Malignant Solid Neoplasm; Refractory Fibrolamellar Carcinoma; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma | interventions — DT2216; Specimen Handling; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DT2216, irinotecan) (Experimental): Patients receive DT2216 IV over 30 minutes on days 1, 4, 8, 11, 15, and 18 of each cycle and irinotecan IV over 90 minutes on days 2-6 of cycle 1, and on days 1-5 of remaining cycles. Cycles repeat every 21 days for up to 35 cycles (24 months) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the trial.
  Interventions: Biological: Bcl-XL Proteolysis Targeting Chimera DT2216; Procedure: Biospecimen Collection; Drug: Irinotecan

INTERVENTIONS:
Biological: Bcl-XL Proteolysis Targeting Chimera DT2216 — Given IV
  Other Names: Antiapoptotic Protein Targeted Degrader DT2216; APTaD DT2216; Bcl-XL Degrader DT2216; Bcl-XL PROTAC DT2216; BCL-XL-specific PROTAC DT2216; DT 2216; DT-2216; DT2216; PROTAC Bcl-XL Deagrader DT2216; PROTAC DT2216; Proteolysis-targeting Chimera Protein Degrader DT2216
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Irinotecan — Given IV

SUMMARY:
This phase I/II trial tests the safety, side effects and best dose of DT2216 in combination with irinotecan and how well it works in treating children, adolescents and young adults with solid tumors and fibrolamellar cancer that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). DT2216 is an anti-apoptotic protein B-cell lymphoma-extra large targeted protein degrader. It may stop the growth of tumor cells by blocking Bcl-xL, a protein needed for tumor cell survival. Irinotecan is in a class of antineoplastic medications called topoisomerase I inhibitors. It blocks a certain enzyme needed for cell division and deoxyribonucleic acid repair and may kill tumor cells. Giving DT2216 in combination with irinotecan may be safe, tolerable, and/or effective in treating children, adolescents and young adults with relapsed or refractory solid tumors or fibrolamellar cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of Bcl-xL proteolysis targeting chimera DT2216 (DT2216) in combination with intravenous irinotecan in patients with recurrent/refractory solid tumors.

II. To define and describe the toxicities of DT2216 in combination with irinotecan administered on this schedule in patients with recurrent/refractory solid tumors and patients with fibrolamellar carcinoma (FLC).

III. To characterize the pharmacokinetics of DT2216 in combination with irinotecan in patients with recurrent/refractory solid tumors and patients with fibrolamellar carcinoma (FLC).

IV. To preliminarily define antitumor activity of DT2216 in combination with irinotecan in patients with recurrent/refractory solid tumors (within the confines of a phase 1 study) and in patients with recurrent/refractory FLC.

SECONDARY OBJECTIVE:

I. To assess the pharmacodynamic activity of DT2216 in combination with irinotecan when administered intravenously in combination to children, adolescents, and young adults with recurrent/refractory cancer (solid tumors and FLC) by measuring peripheral mononuclear cell Bcl-xL levels and, where available, paired pre-treatment and on-(or recently off) treatment tumor samples using immunohistochemistry for TUNEL, Bcl-xL, Bcl2, Mcl1, and Ki67.

EXPLORATORY OBJECTIVES:

I. To explore the correlation of peripheral blood levels of the DNAJB1-PRKACA chimera, vitamin B12 levels and/or a panel of specific genomic markers, as well as intratumoral patterns of infiltrating immune cells as assessed by multiplex immunohistochemistry with disease characteristics of radiographic response in FLC patients.

II. To assess the ability of cross-sectional imaging to identify tumor involved pathological involved (positive) lymph nodes in FLC patients who undergo surgical resection including lymph node sampling or dissection.

OUTLINE: This is a phase I, dose-escalation study of DT2216 in combination with irinotecan, followed by a phase II study.

Patients receive DT2216 intravenously (IV) over 30 minutes on days 1, 4, 8, 11, 15, and 18 of each cycle and irinotecan IV over 90 minutes on days 2-6 of cycle 1, and on days 1-5 of remaining cycles. Cycles repeat every 21 days for up to 35 cycles (24 months) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up every at 3, 6, 9, 12, 18, 24, 36, 48 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* PHASE 1: Patients between ≥ 1 year and ≤ 21 years of age at the time of study enrollment
* PHASE 2: Patients between ≥ 1 year and ≤ 39 years of age at the time of study enrollment
* PHASE 1: Patients with recurrent/refractory solid tumors excluding primary central nervous system tumors
* PHASE 2: Patients with (FLC), which must include genomic confirmation of the DNAJB1:PRKACA fusion performed at a Clinical Laboratory Improvement Act (CLIA)-certified laboratory
* PHASE 1: Patients must have either measurable or evaluable disease
* PHASE 2: Patients must have measurable disease
* PHASE 1: Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* PHASE 2: Patients must have FLC which is recurrent/refractory to at least one line of prior systemic therapy
* Patients with FLC that is unresectable at initial diagnosis but is not recurrent/refractory to at least one prior line of systemic therapy nor metastatic are NOT eligible for either phase 1 or phase 2
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age
* Patients must have fully recovered (grade < 2) from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, eg, blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: See Developmental Therapeutics (DVL) homepage on the Children's Oncology Group (COG) members site for commercial and investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment

    * Solid tumor patients: ≥ 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea). Please refer to the table of myelosuppressive/anticancer agents on the COG website
  * Anti-cancer agents not known to be myelosuppressive (eg, not associated with reduced platelet or absolute neutrophil count [ANC] counts): ≥ 7 days after the last dose of agent. See the DVL homepage on the COG Members site for commercial and investigational agent classifications. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  * Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade ≤ 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: ≥ 14 days after the last dose of a long-acting growth factor (eg, pegfilgrastim) or 7 days for short acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): ≥ 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: ≥ 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: ≥ 30 days
  * Cellular therapy: ≥ 30 days after the completion of any type of cellular therapy (eg, modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiotherapy (XRT)/external beam irradiation including protons: ≥ 14 days after local XRT; ≥ 150 days after TBI, craniospinal XRT or if radiation to ≥ 50% of the pelvis; ≥ 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (eg, radiolabeled antibody, lobenguane I-131 [131I-MIBG]): ≥ 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior Bcl-xL specific therapy (e.g. navitoclax, DT2216). Prior therapy with irinotecan or other topoisomerase 1 inhibitors and/or other BH3 mimetics which are not Bcl-xL selective (e.g. venetoclax) are acceptable
* For patients with solid tumors without known bone marrow involvement: Peripheral absolute neutrophil count (ANC) ≥ 1000/µL
* For patients with solid tumors without known bone marrow involvement: Platelet count ≥ 100,000/µL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity. At least 5 of every cohort of 6 patients must be evaluable for hematologic toxicity for the dose-escalation part of the study. If dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* A creatinine based on age/gender as follows:

  * 1 to < 2 years: Maximum serum creatinine (mg/dL) 0.6 (male), 0.6 (female)
  * 2 to < 6 years: Maximum serum creatinine (mg/dL) 0.8 (male), 0.8 (female)
  * 6 to < 10 years: Maximum serum creatinine (mg/dL) 1 (male), 1 (female)
  * 10 to < 13 years: Maximum serum creatinine (mg/dL) 1.2 (male), 1.2 (female)
  * 13 to < 16 years: Maximum serum creatinine (mg/dL) 1.5 (male), 1.4 (female)
  * 16 to ≤ 39 years: Maximum serum creatinine (mg/dL) 1.7 (male), 1.4 (female)

    * OR a 24 hour urine creatinine clearance ≥ 70 mL/min/1.73 m^2
    * OR a glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard). Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* Patients with solid tumors: Bilirubin (sum of conjugated + unconjugated or total) ≤ 1.5 x upper limit of normal (ULN) for age
* Patients with solid tumors: Alanine aminotransferase (ALT) ≤ 3 x ULN, unless attributed to tumor involvement then ALT ≤ 5 x ULN

  * Note: For the purposes of this study the ULN for ALT is defined as 45 U/L
* Patients with solid tumors: Aspartate aminotransferase (AST) ≤ 3 x ULN, unless attributed to tumor involvement then AST ≤ 5 x ULN

  * Note: For the purposes of this study the ULN for AST is defined as 50 U/L
* Patients with solid tumors: Albumin ≥ 2 g/dL
* Patients with solid tumors: International normalized ratio (INR) ≤ 2.5
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled as evidenced by no increase in seizure frequency in the prior 7 days. If needed, evaluate use of enzyme-inducing anticonvulsants
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5) resulting from prior therapy must be ≤ grade 2, with the exception of decreased tendon reflex (DTR). Patient with any grade of tendon reflex decrease are eligible

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, OR because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (eg, male or female condom) for the duration of the study. Abstinence is an acceptable method of birth control. Patients who could become pregnant should use highly effective contraception during therapy and for 6 months after the last irinotecan dose or 120 days after the last dose of DT2216, whichever is longer. Patients with partners who could become pregnant should use condoms during therapy and for 3 months after the last dose irinotecan or 120 days after the last dose of DT2216, whichever is longer
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who have received drugs that are strong inducers or inhibitors of CYP3A4 within 14 days prior to study enrollment are not eligible
* Patients with lymphoma are excluded
* Patients who have an uncontrolled infection are not eligible
* Patients with grade ≥ 2 diarrhea at baseline are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Dedicated central nervous system (CNS) imaging is not required but patients with current active CNS metastasis whether symptomatic or discovered incidentally without clinical symptoms, are not eligible
* Patients with grade > 2 corrected QT interval (i.e. electrocardiogram [EKG] showing corrected QT interval [QTc] > 480 ms) at baseline are not eligible
* Surgical procedure

  * Central line placement, open or core needle biopsy of sites other than liver: < 2 days prior to enrollment.
  * Open or laparoscopic biopsies or core needle biopsies of liver < 7 days prior to enrollment.
  * All other surgeries < 14 days prior to enrollment

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2031-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study drug
  AEs will be assessed and graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. A descriptive summary of all toxicities will be reported.
Dose-limiting toxicity (DLT) | Up to 21 days
  AEs will be assessed and graded using NCI CTCAE v5.0. A descriptive summary of all toxicities will be reported.
Maximum tolerated dose (MTD)/ recommended phase 2 dose | Up to 21 days
  MTD will be defined as the maximum dose at which fewer than one-third of patients experience DLT during cycle 1 of therapy.
Area under the dose concentration curve of DT2216 | Up to 7 hours
  Median (minimum [min], maximum [max]) area under the dose concentration curve of DT2216 during cycle 1 assessed pre-dose, 5, 30, 60, 180, and 420 minutes post-dose.
Clearance of DT2216 | Up to 7 hours
  Median (min, max) clearance of DT2216 during cycle 1 assessed pre-dose, 5, 30, 60, 180, and 420 minutes post-dose.
Half-life of DT2216 | Up to 7 hours
  Median (min, max) Half-life of DT2216 during cycle 1 assessed pre-dose, 5, 30, 60, 180, and 420 minutes post-dose.
Area under the dose concentration curve of irinotecan | Up to 7 hours
  Median (min, max) area under the dose concentration curve of irinotecan during cycle 1 assessed pre-dose, 5, 30, 60, 180, and 420 minutes post-dose.
Clearance of irinotecan | Up to 7 hours
  Median (min, max) clearance of irinotecan during cycle 1 assessed pre-dose, 5, 30, 60, 180, and 420 minutes post-dose.
Half-life of irinotecan | Up to 7 hours
  Median (min, max) Half-life of irinotecan during cycle 1 assessed pre-dose, 5, 30, 60, 180, and 420 minutes post-dose.
Overall response rate (ORR) | At start of treatment until disease progression or recurrence up to 60 months
  ORR will be recorded from the start of the treatment until disease progression or recurrence. ORR of partial response, complete response or stable disease will be assessed according to Response Evaluation Criteria in Solid Tumors Criteria and will be reported descriptively.

SECONDARY OUTCOMES:
Pharmacodynamic activity | Up to end of cycle 5 (105 days)
  Western blotting will be performed to assess the pharmacodynamic activity by measuring peripheral mononuclear cell Bcl-xL levels.

OTHER OUTCOMES:
Correlation of peripheral blood levels of the DNAJB1-PRKACA chimera | Up to 60 months
  A descriptive analysis of biomarkers will assess associations with disease response. The parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations.
Vitamin B12 levels | Up to 60 months
  A descriptive analysis of biomarkers will assess associations with disease response. The parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations.
Genomic markers panel | Up to 60 months
  Median (interquartile range) ratio of mutant droplet count to total droplet count stratified by study time point.
Intratumoral patterns of infiltrating immune cells | Up to 60 months
  A descriptive analysis of biomarkers will assess associations with disease response. The parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations.
Identification of tumor involved lymph nodes using cross-sectional imaging | Up to 60 months
  Agreement between central pathologic review and central radiology review for relevant resected lymph nodes will be reported using a kappa statistic with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Ortiz, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (19):
- United States (19):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington